CLINICAL TRIAL: NCT01300208
Title: A Phase 2, Pilot, Multicenter, Sequential, Ascending Dose Study to Evaluate the Preliminary Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of CC-11050 in Subjects With Discoid Lupus Erythematosus and Subacute Cutaneous Lupus Erythematosus
Brief Title: To Evaluate the Preliminary Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of CC-11050 in Subjects With Discoid Lupus Erythematosus and Subacute Cutaneous Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-11050-CLE-002
Record Dates: First submitted 2010-10-18; First posted 2011-02-21 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Cutaneous Lupus Erythematosus
Keywords: cutaneous lupus erythematosus; subacute lupus erythematosus; discoid lupus erythematosus; lupus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid | interventions — CC-11050

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): CC-11050 (50 milligrams twice per day and Placebo)
  Interventions: Drug: CC-11050; Other: Placebo
- Cohort 2 (Experimental): CC-11050 (100 milligrams twice per day and Placebo)
  Interventions: Drug: CC-11050; Other: Placebo
- Cohort 3 (Experimental): CC-11050 (200 milligrams twice per day and Placebo)
  Interventions: Drug: CC-11050; Other: Placebo

INTERVENTIONS:
Drug: CC-11050 — Cohort 1: 50 milligrams twice per day for 4 weeks Cohort 2: 100 milligrams twice per day for 8 weeks Cohort 3: 200 milligrams twice per day for 12 week
Other: Placebo

SUMMARY:
This is the first study in cutaneous lupus erythematosus subjects to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and efficacy of CC-11050.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects with a clinical diagnosis of discoid lupus erythematosus or sub acute lupus erythematosus for > 16 weeks prior to screening and consistent histological findings on skin biopsy based on Gilliam classification who are candidates for systemic therapies (as determined by the Investigator)
* Must, in the opinion of the Investigator, have active skin lesions of sufficient severity at Screening and Baseline (a Cutaneous Lupus Area and Severity Index Activity Score of ≥ 10)
* All subjects taking hydroxychloroquine, chloroquine or quinacrine during the study must have documentation of an ophthalmologic exam performed within 24 weeks of the Baseline Visit.
* Must meet the following laboratory criteria:

  * White blood cell count ≥3000/mm3 (≥ 3.0 x 109/L) and < 14,000/mm3 (< 14 x 109/L)
  * Absolute neutrophil count (ANC) > 1500 cells/μL (1.5 x 109/L)
  * Platelet count ≥ 100,000/μL (≥ 100 x 109/L)
  * Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L)
  * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT)
  * ≤ 1.5 X upper limit of normal (ULN)
  * Total bilirubin < 2mg/dL
  * Hemoglobin > 11 g/dL Key Exclusion Criteria
* Participation in multiple CC-11050 cohorts or previous exposure to CC-11050
* Presence or history of SLE based on investigators' clinical evaluation where subject exhibits medically significant (as determined by the Investigator) LE-related pleuritis, pericarditis, neurologic, renal and/or other major SLE-related organ system involvement(SLE-related to SLE joint involvement is acceptable).
* Use of topical or any local therapy known to possibly benefit discoid lupus erythematosus or SCLE sub acute lupus erythematosus within 2 weeks of the Screening Visit
* Use of concomitant disease modifying anti-rheumatic drugs (DMARDs) with the exception of anti-malarials within 4 weeks of screening- Use of topical or any local therapy known to possibly benefit discoid lupus erythematosus or SCLE sub acute lupus erythematosus within 2 weeks of the Screening Visit
* Use of immunosuppressives (eg, azathioprine, mycophenolate mofetil, methotrexate, etc.) within 4 weeks of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2013-03-01 (Actual)

PRIMARY OUTCOMES:
Laboratory values from chemistry, hematology, urinalysis, inflammation/immunology panel that reveal clinically significant abnormalities and that may constitute a safety concern | Up to 21 weeks

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | Up to 21 weeks
  To describe the area under the curve (AUC) of CC-11050 and M15 in plasma
To assess the clinical response rate of CC-11050 in subjects with discoid lupus erythematosus or sub acute lupus erythematosus using the Cutaneous Lupus Area and Severity Index Activity Score following 12-weeks of treatment | 12 weeks
Pharmacokinetics (PK) | Up to 21 weeks
  To describe the peak serum concentration (Cmax) of CC-11050 and M15 in plasma
Pharmacokinetics | Up to 21 weeks
  To describe the lowest serum concentration (Cmin)of CC-11050 and M15 in plasma
Pharmacokinetics (PK) | Up to 21 weeks
  To describe the time after administration of a drug when the maxiumum plasma concentration is reached (tmax) of CC-11050 and M15 in plasma
Pharmacokinetics (PK) | Up to 21 weeks
  To describe the half life (t1/2) of CC-11050 and M15 in plasma
Pharmacokinetics (PK) | Up to 21 weeks
  To describe the oral clearance (CL/F) of CC-11050 and M15 in plasma
Pharmacokinetics (PK) | Up to 21 weeks
  To describe the volume of distribution (Vz/F) of CC-11050 and M15 in plasma

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (19):
- United States (19):
  - Northwest Arkansas Clinical Trials Center, PLLC, Rogers, Arkansas
  - Dermatology Research Associates, Los Angeles, California
  - Medderm Associates, San Diego, California
  - Emory Univ. School of Medicine, Atlanta, Georgia
  - Peachtree Dermatology Associates Research Center, Atlanta, Georgia
  - Central Medaphase Inc, Newnan, Georgia
  - Northwestern University, Chicago, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - DermResearch, PLLC, Louisville, Kentucky
  - Dermatology & Advanced Aesthetics, Lake Charles, Louisiana
  - Central Dermatology, P.C., St Louis, Missouri
  - NYU Langone Medical Center, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Penn State Hershey Dermatology, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - UT Southwestern Medical Center Dallas, Dallas, Texas